CLINICAL TRIAL: NCT01384734
Title: A Phase IIb Randomized, Controlled, Partially-Blinded Trial to Investigate Safety, Efficacy and Dose-Response of BMS-663068 in Treatment-experienced HIV-1 Subjects, Followed by an Open-Label Period on the Recommended Dose
Brief Title: HIV Attachment Inhibitor to Treat Human Immunodeficiency Virus 1 (HIV-1) Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 205889; AI438-011 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2011-06-23; First posted 2011-06-29 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-08

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir; Raltegravir Potassium; Tenofovir; Ritonavir; Atazanavir Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm A: BMS-663068 (400mg) + Raltegravir + Tenofovir (Experimental): Treatment Group 1
  Interventions: Drug: BMS-663068 400 mg; Drug: Raltegravir 400 mg; Drug: Tenofovir 300 mg
- Arm B: BMS-663068 (800 mg) + Raltegravir + Tenofovir (Experimental): Treatment Group 2
  Interventions: Drug: BMS-663068 800 mg; Drug: Raltegravir 400 mg; Drug: Tenofovir 300 mg
- Arm C: BMS-663068 (600 mg) + Raltegravir + Tenofovir (Experimental): Treatment Group 3
  Interventions: Drug: BMS-663068 600 mg; Drug: Raltegravir 400 mg; Drug: Tenofovir 300 mg
- Arm D: BMS-663068 (1200 mg) + Raltegravir + Tenofovir (Experimental): Treatment Group 4
  Interventions: Drug: BMS-663068 1200 mg; Drug: Raltegravir 400 mg; Drug: Tenofovir 300 mg
- Arm E: Atazanavir + Ritonavir + Raltegravir + Tenofovir (Active Comparator): Treatment Group 1 (reference arm)
  Interventions: Drug: Raltegravir 400 mg; Drug: Tenofovir 300 mg; Drug: Ritonavir 100 mg; Drug: Atazanavir 300 mg

INTERVENTIONS:
Drug: BMS-663068 400 mg — Tablets, Oral, 400 mg, twice daily (BID), 24+ weeks until optimal dose is selected, or 96 weeks if optimal dose
  Arms: Arm A: BMS-663068 (400mg) + Raltegravir + Tenofovir
Drug: BMS-663068 800 mg — Tablets, Oral, 800 mg, twice daily (BID), 24+ weeks until optimal dose is selected, or 96 weeks if optimal dose
  Arms: Arm B: BMS-663068 (800 mg) + Raltegravir + Tenofovir
Drug: BMS-663068 600 mg — Tablets, Oral, 600 mg, once daily (QD), 24+ weeks until optimal dose is selected, or 96 weeks if optimal dose
  Arms: Arm C: BMS-663068 (600 mg) + Raltegravir + Tenofovir
Drug: BMS-663068 1200 mg — Tablets, Oral, 1200 mg, once daily (QD), 24+ weeks until optimal dose is selected, or 96 weeks if optimal dose
  Arms: Arm D: BMS-663068 (1200 mg) + Raltegravir + Tenofovir
Drug: Raltegravir 400 mg — Tablets, Oral, 400 mg, twice daily (BID), 24+ weeks until optimal dose is selected, or 96 weeks if optimal dose
Drug: Tenofovir 300 mg — Tablets, Oral, 300 mg, Once daily (QD), 24+ weeks until optimal dose is selected, or 96 weeks if optimal dose
Drug: Ritonavir 100 mg — Tablets, Oral, 100 mg, Once daily, 96 weeks
  Arms: Arm E: Atazanavir + Ritonavir + Raltegravir + Tenofovir
Drug: Atazanavir 300 mg — Capsules, Oral, 300 mg, Once daily, 96 weeks
  Arms: Arm E: Atazanavir + Ritonavir + Raltegravir + Tenofovir

SUMMARY:
The purpose of this study is to assess the safety, efficacy, tolerability and pharmacokinetics of four doses of BMS-663068 with Raltegravir (RAL) + Tenofovir Disoproxil Fumarate (TDF). At least 1 dose of BMS-663068 can be identified which is safe, well tolerated, and efficacious when combined with RAL + TDF for treatment-experienced HIV-1 infected subjects. PHENOSENSE® is a registered trademark of Monogram Biosciences.

DETAILED DESCRIPTION:
Masking: Double-blind for BMS-6630368 treatment groups until the Week 24 Primary Endpoint analysis, then open label. The reference groups is all open-label.

Arms: 5 (4 BMS-663068 treatment groups and 1 reference group)

Intervention Model: Parallel (with unblinding after the Week 24 primary endpoint analysis)

ELIGIBILITY:
Inclusion Criteria:

* Plasma HIV-1 RNA ≥ 1000 copies/ml at Screening
* Treatment experience with antiretroviral therapies (excluding integrase inhibitors)
* Screening PHENOSENSE Entry indicating BMS-626529 inhibitory concentration (IC)50 < 0.1 μM
* Cluster of differentiation (CD)4+ T-cell count > 50 cells/mm3

Exclusion Criteria:

* History (or evidence at Screening) of genotypic resistance to any component of the study regimen [ Tenofovir Disoproxil Fumarate (TDF), Atazanavir (ATV), Raltegravir (RAL)]
* Certain laboratory and electrocardiogram (ECG) values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2011-07-26 (Actual); Primary Completion 2013-02-18 (Actual); Study Completion 2017-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (45):
- United States (12):
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Longview, Texas
- Argentina (5):
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Rosario
- GSK Investigational Site, Bogotá, Colombia
- Germany (4):
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, München
- Mexico (7):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, San Luis Potosí City, San Luis Potosí
  - GSK Investigational Site, Aguascalientes
  - GSK Investigational Site, DF
  - GSK Investigational Site, Distrito Federal
  - GSK Investigational Site, Mexico City
- Peru (2):
  - GSK Investigational Site, Iquitos, Loreto
  - GSK Investigational Site, Lima
- Romania (4):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Iași
- Russia (2):
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
- South Africa (4):
  - GSK Investigational Site, Dundee, KwaZulu-Natal
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Observatory, Cape Town
- Spain (4):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Madrid

REFERENCES:
- [Derived] Thompson M, Lalezari JP, Kaplan R, Pinedo Y, Pena OAS, Cahn P, Stock DA, Joshi SR, Hanna GJ, Lataillade M; AI438011 study team. Safety and efficacy of the HIV-1 attachment inhibitor prodrug fostemsavir in antiretroviral-experienced subjects: week 48 analysis of AI438011, a Phase IIb, randomized controlled trial. Antivir Ther. 2017;22(3):215-223. doi: 10.3851/IMP3112. Epub 2016 Dec 6. PMID 27922453
- [Derived] Landry I, Zhu L, Abu Tarif M, Hruska M, Sadler BM, Pitsiu M, Joshi S, Hanna GJ, Lataillade M, Boulton DW, Bertz RJ. Model-Based Phase 3 Dose Selection for HIV-1 Attachment Inhibitor Prodrug BMS-663068 in HIV-1-Infected Patients: Population Pharmacokinetics/Pharmacodynamics of the Active Moiety, BMS-626529. Antimicrob Agents Chemother. 2016 Apr 22;60(5):2782-9. doi: 10.1128/AAC.02503-15. Print 2016 May. PMID 26902761
- [Derived] Lalezari JP, Latiff GH, Brinson C, Echevarria J, Trevino-Perez S, Bogner JR, Thompson M, Fourie J, Sussmann Pena OA, Mendo Urbina FC, Martins M, Diaconescu IG, Stock DA, Joshi SR, Hanna GJ, Lataillade M; AI438011 study team. Safety and efficacy of the HIV-1 attachment inhibitor prodrug BMS-663068 in treatment-experienced individuals: 24 week results of AI438011, a phase 2b, randomised controlled trial. Lancet HIV. 2015 Oct;2(10):e427-37. doi: 10.1016/S2352-3018(15)00177-0. Epub 2015 Sep 1. PMID 26423650
- [Derived] Zhou N, Nowicka-Sans B, McAuliffe B, Ray N, Eggers B, Fang H, Fan L, Healy M, Langley DR, Hwang C, Lataillade M, Hanna GJ, Krystal M. Genotypic correlates of susceptibility to HIV-1 attachment inhibitor BMS-626529, the active agent of the prodrug BMS-663068. J Antimicrob Chemother. 2014 Mar;69(3):573-81. doi: 10.1093/jac/dkt412. Epub 2013 Oct 14. PMID 24128669

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Human Immunodeficiency Virus (HIV-1) were randomized in ratio of 1:1:1:1:1 to 5 treatment arms of the study. Four groups with distinct dose of Fostemsavir (FTR, also referred BMS-663068) with Raltegravir (RAL) Tenofovir Disoproxil Fumarate (TDF). There was a reference group with ritonavir (r) boosted atazanavir (ATV), RAL and TDF.
Pre-assignment Details: A total of 581 participants were screened, 254 were enrolled of which 2 participants withdrew consent and 1 was randomized in error. A total 251 participants were randomized and treated of which 32 were in Monotherapy sub-study (only FTR) and continued to Primary study.
Groups:
- FTR 400 mg BID/RAL/TDF: Participants were randomized and administered 400 milligrams (mg) FTR twice daily (BID) (double-blind) along with 400 mg RAL BID (open label) and 300 mg TDF once daily (QD) (open label).
- FTR 800 mg BID/RAL/TDF: Participants were randomized and administered 800 mg of FTR BID (double-blind) along with 400 mg RAL BID (open label) and 300 mg TDF QD (open label).
- FTR 600 mg QD/RAL/TDF: Participants were randomized and administered 600 mg of FTR QD (double-blind) along with 400 mg RAL BID (open label) and 300 mg TDF QD (open label).
- FTR 1200 mg QD/RAL/TDF: Participants were randomized and administered 1200 mg of FTR QD along (double-blind) with 400 mg RAL BID (open label) and 300 mg TDF QD (open label).
- ATV/r/RAL/TDF: Participants were randomized to Reference group (open label) and administered ATV/r 300/100 mg once daily along with 400 mg RAL BID and 300 mg TDF QD.
Period: Overall Study
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF | ATV/r/RAL/TDF
Started | 50 | 49 | 51 | 50 | 51
Completed | 33 | 25 | 28 | 22 | 22
Not Completed | 17 | 24 | 23 | 28 | 29
Not completed — Adverse Event | 0 | 3 | 0 | 2 | 7
Not completed — Death | 1 | 0 | 1 | 0 | 0
Not completed — Continuation criteria not met | 0 | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 3 | 7 | 4 | 4 | 2
Not completed — Lost to Follow-up | 5 | 3 | 3 | 8 | 5
Not completed — Non-compliance with study drug | 1 | 2 | 6 | 0 | 2
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 1
Not completed — Sponsor terminated | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 5 | 6 | 7 | 9
Not completed — Investigator relocating | 0 | 2 | 0 | 3 | 1
Not completed — Unable to come back for visit | 1 | 0 | 1 | 1 | 0
Not completed — Prison | 0 | 0 | 1 | 0 | 0
Not completed — As per Exclusion criteria | 0 | 1 | 0 | 0 | 0
Not completed — Missed End of treatment visit | 0 | 0 | 0 | 1 | 0
Not completed — Adhesion problem | 0 | 0 | 0 | 1 | 0
Not completed — Early termination | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FTR 400 mg BID/RAL/TDF: Participants were randomized and administered 400 mg FTR BID (double-blind) along with 400 mg RAL BID (open label) and 300 mg TDF once daily (QD) (open label).
- Total: Total of all reporting groups
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF | ATV/r/RAL/TDF | Total
Number analyzed (Participants) | 50 | 49 | 51 | 50 | 51 | 251
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (8.17) | 38.4 (9.49) | 40.1 (9.45) | 39.2 (11.41) | 39.7 (10.63) | 39.1 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 22 | 16 | 22 | 100
  Male | 31 | 28 | 29 | 34 | 29 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 14 | 15 | 16 | 18 | 13 | 76
  American Indian Or Alaska Native | 0 | 0 | 1 | 1 | 1 | 3
  Asian | 0 | 2 | 0 | 0 | 0 | 2
  White | 20 | 19 | 17 | 16 | 23 | 95
  Other/Mixed | 16 | 13 | 17 | 15 | 14 | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) < 50 Copies Per Milliliter (c/mL) at Week 24
Description: Percentage of participants with plasma HIV 1 RNA < 50 c/mL at Week 24 using the Food and Drug Administration (FDA) snapshot algorithm was assessed to evaluate the antiviral activity. Treatment comparisons were not performed as this was an estimation study. Response rates were tabulated by treatment arm with exact Clopper-Pearson binomial 95 percentage confidence intervals (CI). Virologic success or failure was determined by the last available HIV-1 RNA assessment while the participant was on-treatment within the snapshot window of the visit of interest. Intent-To-Treat-Exposed (ITT-E) Population includes all randomized participants who received at least one dose of study treatment.
Time Frame: Week 24
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF | ATV/r/RAL/TDF
Number analyzed (Participants) | 50 | 49 | 51 | 50 | 51
Percentage of Participants | 80 [66.3 to 90.0] | 69 [54.6 to 81.7] | 76 [62.5 to 87.2] | 72 [57.5 to 83.8] | 75 [60.4 to 85.7]

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAE) and Discontinuation Due to AEs up to Week 24
Description: Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or suspected transmission of an infectious agent via the study drug were categorized as SAE. AEs leading to discontinuation of study therapy were also reported as safety assessment. Safety population included all participants who received at least one dose of study treatment. Summaries of SAEs and AEs leading to discontinuation or withdrawal through Week 24 included AEs with onset on or after the start of study treatment (i.e. study date of first study treatment intake) up to and including the end of the Week 24 visit snapshot window.
Time Frame: Up to Week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF | ATV/r/RAL/TDF
Number analyzed (Participants) | 50 | 49 | 51 | 50 | 51
Participants
  SAE | 3 | 4 | 4 | 2 | 5
  AEs leading to discontinuation | 1 | 2 | 0 | 1 | 2

3. Secondary Outcome: Change From Monotherapy Baseline in log10 HIV RNA of the Monotherapy Period
Description: Change from monotherapy Baseline in log10 HIV RNA to assess the antiviral activity of temsavir following administration of selected doses of FTR administered orally to HIV-1-infected participants for 7 days. Baseline is defined as the last non-missing value on or before the date of first dose of study treatment. Change from Baseline was calculated as value at indicated time point minus Baseline value. ITT-E Monotherapy Population comprised of participants that were randomized and participated in the monotherapy sub-study and received at least one dose of FTR Monotherapy. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to Day 8 of the monotherapy period
Population: ITT-E Monotherapy Population
Measure: Mean (Standard Deviation); unit: log10 c/mL
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF
Number analyzed (Participants) | 7 | 5 | 10 | 10
log10 c/mL
  Day 2, n=7, 5, 10, 9: number analyzed (Participants) | 7 | 5 | 10 | 9
  Day 2, n=7, 5, 10, 9 | 0.220 (0.1630) | 0.149 (0.1820) | 0.126 (0.1811) | 0.126 (0.4216)
  Day 5, n=7, 4, 10, 10: number analyzed (Participants) | 7 | 4 | 10 | 10
  Day 5, n=7, 4, 10, 10 | -0.340 (0.3185) | -0.811 (0.3455) | -0.593 (0.2429) | -0.767 (0.6388)
  Day 6, n=7, 5, 10, 10 | -0.530 (0.3170) | -1.082 (0.3388) | -0.822 (0.3076) | -1.053 (0.7491)
  Day 7, n=6, 5, 10, 10: number analyzed (Participants) | 6 | 5 | 10 | 10
  Day 7, n=6, 5, 10, 10 | -0.556 (0.4264) | -1.443 (0.4484) | -1.086 (0.4216) | -1.198 (0.6863)
  Day 8, n=6, 4, 9, 9: number analyzed (Participants) | 6 | 4 | 9 | 9
  Day 8, n=6, 4, 9, 9 | -0.691 (0.5380) | -1.372 (0.3208) | -1.218 (0.3902) | -1.470 (0.6570)

4. Secondary Outcome: Maximum Decrease From Monotherapy Baseline in log10 Plasma HIV-1 RNA
Description: Maximum decrease from monotherapy Baseline in log10 plasma HIV-1 RNA during monotherapy to assess the antiviral activity of temsavir following administration of selected doses of FTR administered orally to HIV-1-infected participants for 7 days. Baseline is defined as the last non-missing value on or before the date of first dose of study treatment. Change from Baseline was calculated as value at indicated time point minus Baseline value. The data for monotherapy nadir has been presented where nadir represents the maximum decrease from Baseline.
Time Frame: Baseline and up to Day 8 of the monotherapy period
Population: ITT-E Monotherapy Population
Measure: Mean (Standard Deviation); unit: log10 c/mL
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF
Number analyzed (Participants) | 7 | 5 | 10 | 10
log10 c/mL | -0.770 (0.4487) | -1.524 (0.3898) | -1.250 (0.3818) | -1.399 (0.6688)

5. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA < 50 c/mL at Day 8 of the Monotherapy Period
Description: Percentage of participants with plasma HIV 1 RNA < 50 c/mL at Baseline of combination therapy was assessed to evaluate the antiviral activity of four doses of FTR. Baseline of combination therapy was the Day 1 of the combination therapy. Virologic success or failure was determined using the non-missing viral load value at Baseline of combination therapy. The assessment closest to the window target Study Day was used for the analysis. Only those participants with data available at the specified time points were analyzed.
Time Frame: Up to Day 8 of the monotherapy period
Population: ITT-E Monotherapy Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF
Number analyzed (Participants) | 6 | 4 | 9 | 9
Percentage of Participants | 0 [0.0 to 45.9] | 0 [0.0 to 60.2] | 0 [0.0 to 33.6] | 11 [0.3 to 48.2]

6. Secondary Outcome: Number of Participants With SAE and Discontinuation Due to AEs During Monotherapy Period
Description: Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or suspected transmission of an infectious agent via the study drug were categorized as SAE. AEs leading to discontinuation of study therapy were also reported as safety assessment.
Time Frame: Up to Day 8 of the monotherapy period
Population: ITT-E Monotherapy Population
Measure: Count of Participants; unit: Participants
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF
Number analyzed (Participants) | 7 | 5 | 10 | 10
Participants
  SAE | 0 | 0 | 0 | 0
  AEs leading to discontinuation | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Monotherapy Baseline in Cluster of Differentiation (CD)4+ and CD8+ T-cell Counts During Monotherapy
Description: Blood was collected and CD4+ and CD8+ cell count assessment was done by flow cytometery and was carried out at Baseline (Day 1) to evaluate the immunological activity of multiple doses of FTR. Baseline is defined as the last non-missing value on or before the date of first dose of study treatment and the values are absolute values. Change from Baseline was calculated as value at indicated time point minus Baseline value. Only those participants with data available at the specified time points were analyzed.
Time Frame: Baseline and Day 8
Population: ITT-E Monotherapy Population
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF
Number analyzed (Participants) | 5 | 4 | 8 | 8
cells per cubic millimeter
  CD4+ | 58.4 (81.60) | 134.8 (25.70) | 71.8 (117.68) | 63.4 (100.86)
  CD8+ | 134.2 (180.64) | 216.3 (215.57) | 188.0 (363.58) | 67.6 (236.55)

8. Secondary Outcome: Change From Monotherapy Baseline in CD4+ and CD8+ T-cell Proportion During Monotherapy
Description: Blood was collected and CD4+ and CD8+ proportion assessment was done by flow cytometery and was carried out at Baseline (Day 1) to evaluate the immunological activity of multiple doses of FTR. Baseline is defined as the last non-missing value on or before the date of first dose of study treatment and the values are absolute values. Change from Baseline was calculated as value at indicated time point minus Baseline value. Only those participants with data available at the specified time points were analyzed.
Time Frame: Baseline and Day 8
Population: ITT-E Monotherapy Population
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF
Number analyzed (Participants) | 6 | 4 | 9 | 8
cells per cubic millimeter
  CD4+ | -0.005 (0.0084) | 0.023 (0.0299) | 0.008 (0.0335) | 0.014 (0.0320)
  CD8+ | -0.003 (0.0273) | -0.040 (0.0245) | -0.009 (0.0465) | -0.021 (0.0364)

9. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA < 50 c/mL at Primary Study
Description: Percentage of participants with plasma HIV 1 RNA < 50 c/mL at Weeks 48 and 96 using the FDA snapshot algorithm was assessed to evaluate the antiviral activity. Treatment comparisons were not performed as this was an estimation study. Response rates were tabulated by treatment arm with exact Clopper-Pearson binomial 95 percentage CI. Virologic success or failure was determined by the last available HIV-1 RNA assessment while the participant was on-treatment within the snapshot window of the visit of interest.
Time Frame: Weeks 48 and 96
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF | ATV/r/RAL/TDF
Number analyzed (Participants) | 50 | 49 | 51 | 50 | 51
Percentage of Participants
  Week 48 | 82 [68.6 to 91.4] | 61 [46.2 to 74.8] | 69 [54.1 to 80.9] | 68 [53.3 to 80.5] | 71 [56.2 to 82.5]
  Week 96 | 78 [64.0 to 88.5] | 49 [34.4 to 63.7] | 63 [48.1 to 75.9] | 58 [43.2 to 71.8] | 57 [42.2 to 70.7]

10. Secondary Outcome: Number of Participants With SAE and Discontinuation Due to AEs During Primary Study
Description: Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or suspected transmission of an infectious agent via the study drug were categorized as SAE. AEs leading to discontinuation of study therapy were also reported as safety assessment. Safety Population comprised of participants who received at least one dose of study treatment. Summaries of SAEs and AEs leading to discontinuation or withdrawal through Week X (where X = 48 or 96) included AEs with onset on or after the start of study treatment (i.e. study date of first study treatment intake) up to and including the end of the Week 48 and 96 visit snapshot window.
Time Frame: Weeks 48 and 96
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF | ATV/r/RAL/TDF
Number analyzed (Participants) | 50 | 49 | 51 | 50 | 51
Participants
  SAE, Week 48 | 3 | 5 | 4 | 2 | 5
  SAE, Week 96 | 5 | 7 | 6 | 4 | 7
  AEs leading to discontinuation, Week 48 | 1 | 2 | 0 | 1 | 3
  AEs leading to discontinuation, Week 96 | 1 | 2 | 0 | 2 | 5

11. Secondary Outcome: Change From Baseline in CD4+ T-cell Count
Description: Blood was collected and CD4+ cell count assessment by flow cytometery was carried out at Baseline (Day 1), Weeks 24, 48 and 96 to evaluate the immunological activity of multiple doses of BMS-663068/GSK3684934. Baseline is defined as the last non-missing value on or before the date of first dose of study treatment and those values are absolute values. Change from Baseline was calculated as value at indicated time point minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 24, 48 and 96
Population: ITT-E Population
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF | ATV/r/RAL/TDF
Number analyzed (Participants) | 50 | 49 | 51 | 50 | 51
Cells per cubic millimeter
  Week 24, n=41, 38, 48, 42, 40: number analyzed (Participants) | 41 | 38 | 48 | 42 | 40
  Week 24, n=41, 38, 48, 42, 40 | 134.3 (84.63) | 111.0 (123.75) | 109.5 (87.20) | 124.5 (111.04) | 119.4 (142.85)
  Week 48, n=43, 34, 43, 41, 41: number analyzed (Participants) | 43 | 34 | 43 | 41 | 41
  Week 48, n=43, 34, 43, 41, 41 | 199.1 (124.24) | 158.7 (118.70) | 140.5 (97.16) | 155.4 (107.06) | 178.7 (133.90)
  Week 96, n=42, 28, 35, 28, 31: number analyzed (Participants) | 42 | 28 | 35 | 28 | 31
  Week 96, n=42, 28, 35, 28, 31 | 264.6 (147.83) | 210.8 (158.03) | 175.7 (98.28) | 211.7 (151.03) | 250.1 (217.54)

12. Secondary Outcome: Number of Participants With Newly-emergent Genotypic Substitutions at Week 24
Description: Participants who administered antiretroviral (ARV) with virologic failure (VF) were assessed. Genotypic substitution included assessment of Reverse Transcriptase (RT) substitution, Protease Inhibitor (PI) substitution and Integrase RAL substitution as per International Acquired Immune Deficiency Syndrome (AIDS) Society-USA (IAS-USA) list. ITT-E Resistance Tested through Week 24 population included participants who met the criteria for Resistance testing, and the confirmatory value or value at discontinuation occurred at or before the end of the Week 24 Snapshot analysis window. The criteria for resistance tested was participant who had virologic failure or met the following criteria a) Participants who achieved viral suppression (plasma HIV-1 RNA < 50 c/mL) and have confirmed plasma HIV-1 RNA >= 400 c/mL at any time during the study. b) Participants who were discontinued before achieving viral suppression (plasma HIV-1 RNA < 50 c/mL) after Week 8 with last plasma HIV-1 RNA >=400 c/mL.
Time Frame: Up to Week 24
Population: ITT-E Resistance Tested through Week 24 Population
Measure: Count of Participants; unit: Participants
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF | ATV/r/RAL/TDF
Number analyzed (Participants) | 3 | 7 | 11 | 3 | 5
Participants
  PI substitution | 0 | 0 | 0 | 0 | 0
  RT substitution | 0 | 0 | 0 | 1 | 0
  Integrase substitution | 0 | 0 | 1 | 1 | 0

13. Secondary Outcome: Number of Participants With Newly-emergent Genotypic Substitutions at Week 48
Description: Participants who administered ARV with VF were assessed. Genotypic substitution included assessment of RT substitution, PI substitution and Integrase RAL substitution as per IAS-USA list. ITT-E Resistance Tested through Week 48 population included participants who met the criteria for Resistance testing, and the confirmatory value or value at discontinuation occurred at or before the end of the Week 48 Snapshot analysis window. The criteria for resistance tested was participant who had virologic failure or the following criteria a) Participants who achieved viral suppression (plasma HIV-1 RNA < 50 c/mL) and have confirmed plasma HIV-1 RNA >= 400 c/mL at any time during the study. b) Participants who were discontinued before achieving viral suppression (plasma HIV-1 RNA < 50 c/mL) after Week 8 with last plasma HIV-1 RNA >=400 c/mL.
Time Frame: Up to Week 48
Population: ITT-E Resistance Tested through Week 48 Population
Measure: Count of Participants; unit: Participants
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF | ATV/r/RAL/TDF
Number analyzed (Participants) | 9 | 10 | 16 | 9 | 6
Participants
  PI substitution | 1 | 0 | 0 | 1 | 0
  RT substitution | 0 | 0 | 0 | 2 | 0
  Integrase substitution | 1 | 1 | 1 | 2 | 0

14. Secondary Outcome: Number of Participants With Newly-emergent Genotypic Substitutions at Week 96
Description: Participants who administered ARV with VF were assessed. Genotypic substitution included assessment of RT substitution, PI substitution and Integrase RAL substitution as per IAS-USA list. ITT-E Resistance Tested through Week 96 population included participants who met the criteria for Resistance testing, and the confirmatory value or value at discontinuation occurred at or before the end of the Week 96 Snapshot analysis window. The criteria for resistance tested was participants with virologic failure or the following criteria a) Participants who achieved viral suppression (plasma HIV-1 RNA < 50 c/mL) and have confirmed plasma HIV-1 RNA >= 400 c/mL at any time during the study. b) Participants who were discontinued before achieving viral suppression (plasma HIV-1 RNA < 50 c/mL) after Week 8 with last plasma HIV-1 RNA >=400 c/mL.
Time Frame: Up to Week 96
Population: ITT-E Resistance Tested through Week 96 Population
Measure: Count of Participants; unit: Participants
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF | ATV/r/RAL/TDF
Number analyzed (Participants) | 20 | 18 | 23 | 13 | 11
Participants
  PI substitution | 3 | 1 | 2 | 2 | 0
  RT substitution | 2 | 1 | 2 | 2 | 1
  Integrase RAL substitution | 2 | 2 | 1 | 3 | 0

15. Secondary Outcome: Maximum Change From Baseline in Inhibitory Concentration at 50% (IC50) Fold Change Among Participants With VF at Week 24
Description: Virologic failure is defined clinically as confirmed plasma HIV-1 RNA >= 50 copies/mL at Week 24 or later or virologic rebound defined as confirmed HIV-1 RNA >=50 copies/mL at any time after prior confirmed suppression to <50 copies/mL OR confirmed >1 log10 copies/mL increase in HIV-1 RNA at any time above nadir level where nadir was >= 50 copies/mL . The phenotypic resistance to a drug is defined as a fold change (i.e, ratio of the IC50 of the clinical isolate to the IC50 of the reference strain) greater than the cut-off for reduced susceptibility. Maximum change from Baseline in Temsavir IC50 fold change based on all on-treatment values has been presented. Baseline is defined as the last non-missing value on or before the date of first dose of study treatment and those values are absolute values. Change from Baseline was calculated as value at indicated time point minus Baseline value. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline and up to Week 24
Population: ITT-E Resistance Tested through Week 24 Population
Measure: Mean (Standard Deviation); unit: IC50 Fold Change
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF
Number analyzed (Participants) | 3 | 4 | 6 | 2
IC50 Fold Change | -2.350 (3.4536) | 1014.748 (2015.5876) | 101.627 (190.4849) | 39.030 (55.1119)

16. Secondary Outcome: Change From Baseline in IC50 Fold Change Among Participants With VF at Week 48
Description: Virologic failure is defined clinically as confirmed plasma HIV-1 RNA >= 50 copies/mL at Week 24 or later or later or virologic rebound defined as confirmed HIV-1 RNA >=50 copies/mL at any time after prior confirmed suppression to <50 copies/mL OR confirmed >1 log10 copies/mL increase in HIV-1 RNA at any time above nadir level where nadir was >= 50 copies/mL. The phenotypic resistance to a drug is defined as a fold change (i.e, ratio of the IC50 of the clinical isolate to the IC50 of the reference strain) greater than the cut-off for reduced susceptibility. Maximum change from Baseline in Temsavir IC50 fold change based on all on-treatment values has been presented. Baseline is defined as the last non-missing value on or before the date of first dose of study treatment and those values are absolute values. Change from Baseline was calculated as value at indicated time point minus Baseline value. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline and up to Week 48
Population: ITT-E Resistance Tested through Week 48 Population
Measure: Mean (Standard Deviation); unit: IC50 Fold Change
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF
Number analyzed (Participants) | 5 | 7 | 8 | 5
IC50 Fold Change | -2.624 (3.2819) | 586.776 (1521.9126) | 81.729 (165.4931) | 449.092 (647.9828)

17. Secondary Outcome: Change From Baseline in IC50 Fold Change Among Participants With VF at Week 96
Description: Virologic failure is defined clinically as confirmed plasma HIV-1 RNA >= 50 copies/mL at Week 24 or later or virologic rebound defined as confirmed HIV-1 RNA >=50 copies/mL at any time after prior confirmed suppression to <50 copies/mL OR confirmed >1 log10 copies/mL increase in HIV-1 RNA at any time above nadir level where nadir was >= 50 copies/mL. The phenotypic resistance to a drug is defined as a fold change (i.e, ratio of the IC50 of the clinical isolate to the IC50 of the reference strain) greater than the cut-off for reduced susceptibility. Maximum change from Baseline in Temsavir IC50 fold change based on all on-treatment values has been presented. Baseline is defined as the last non-missing value on or before the date of first dose of study treatment and those values are absolute values. Change from Baseline was calculated as value at indicated time point minus Baseline value. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline and up to Week 96
Population: ITT-E Resistance Tested through Week 96 Population
Measure: Mean (Standard Deviation); unit: IC50 Fold Change
Arm/Group | FTR 400 mg BID/RAL/TDF | FTR 800 mg BID/RAL/TDF | FTR 600 mg QD/RAL/TDF | FTR 1200 mg QD/RAL/TDF
Number analyzed (Participants) | 6 | 14 | 11 | 9
IC50 Fold Change | 25.480 (68.9030) | 419.901 (1092.5929) | 46.351 (157.9219) | 777.818 (1550.8887)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of study treatment (Day 1) until 2117 days
Description: The analysis was based on the Safety Population. Adverse events data were not reported cumulatively for all intervention concentrations, and were only reported cumulatively per FTR or ATV/r interventions.
Groups:
- FTR/RAL/TDF Total: All participants who were randomized to receive either of FTR 400mg BID, 800 mg BID, 600mg QD or 1200 mg QD (double-blind) along with 400 mg RAL BID (open label) and 300 mg TDF QD (open label).
Arm/Group | FTR/RAL/TDF Total | ATV/r/RAL/TDF
All-Cause Mortality (participants affected / at risk) | 3/200 | 0/51
Serious Adverse Events (participants affected / at risk) | 35/200 | 8/51
Other Adverse Events (participants affected / at risk) | 163/200 | 46/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FTR/RAL/TDF Total (N=200) | ATV/r/RAL/TDF (N=51)
Bone tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 3 (5) | 1 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Adenocarcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FTR/RAL/TDF Total (N=200) | ATV/r/RAL/TDF (N=51)
Nasopharyngitis (Infections and infestations) | 32 (52) | 5 (10)
Upper respiratory tract infection (Infections and infestations) | 27 (47) | 7 (7)
Urinary tract infection (Infections and infestations) | 28 (62) | 6 (19)
Influenza (Infections and infestations) | 22 (43) | 7 (8)
Bronchitis (Infections and infestations) | 22 (34) | 4 (4)
Pharyngitis (Infections and infestations) | 17 (19) | 5 (5)
Herpes zoster (Infections and infestations) | 17 (20) | 2 (2)
Gastroenteritis (Infections and infestations) | 11 (11) | 6 (6)
Lower respiratory tract infection (Infections and infestations) | 10 (12) | 1 (1)
Onychomycosis (Infections and infestations) | 8 (8) | 3 (3)
Sinusitis (Infections and infestations) | 5 (12) | 4 (12)
Diarrhoea (Gastrointestinal disorders) | 37 (48) | 10 (16)
Nausea (Gastrointestinal disorders) | 19 (22) | 6 (18)
Vomiting (Gastrointestinal disorders) | 16 (18) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 13 (13) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 12 (13) | 2 (2)
Constipation (Gastrointestinal disorders) | 11 (12) | 0 (0)
Headache (Nervous system disorders) | 38 (64) | 6 (18)
Dizziness (Nervous system disorders) | 9 (9) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (25) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (22) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (17) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 9 (16) | 3 (5)
Alanine aminotransferase increased (Investigations) | 6 (6) | 4 (6)
Blood bilirubin increased (Investigations) | 1 (1) | 4 (9)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 11 (35)
Jaundice (Hepatobiliary disorders) | 0 (0) | 8 (9)
Ocular icterus (Hepatobiliary disorders) | 1 (1) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 15 (21) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 15 (16) | 3 (3)
Fatigue (General disorders) | 11 (14) | 4 (4)
Insomnia (Psychiatric disorders) | 13 (16) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.